CLINICAL TRIAL: NCT06273358
Title: The Effect of Preoperative Sleep Quality on Postoperative Delirium Status in Adult Patients
Brief Title: Preoperative Sleep Quality and Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Yasin Tire, MD, Assoc. Prof. Dr. Yasin Tire, Konya City Hospital
Other Study IDs: Study Sleep Quality
Record Dates: First submitted 2023-12-14; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: PREOPERATIVE SLEEP QUALITY ON POSTOPERATIVE DELIRIUM
Keywords: General anesthesia; Delirium; Perioperative neurocognitive disorders; Sleep Quality
MeSH Terms: conditions — Delirium; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Over 45 year old: Before surgery All preoperative patients will have Preoperative Stop Bang, Pittsburghb Sleep Quality Index, and Mini Mental tests for sleep quality and consciousness monitoring. This will be based on sleep the day before surgery and mini-mental exams before surgery.
  The intraoperative phase Our clinical approach is to admit patients under general anesthesia after regular assessment and monitoring. The following parameters will be recorded intraoperatively.
  After surgery As usual, patients are brought to the PACU after awakening. It will be measured Pittsburghb Sleep Quality Index on 3 days, QoR-15 on the last day, and 3D CAM or ICU-CAM for 3 days postoperatively. Patients will stay in the ward and intensive care unit for 72 hours and be called for 72 hours after release.
- Over 65 year old: Before surgery All preoperative patients will have Preoperative Stop Bang, Pittsburghb Sleep Quality Index, and Mini Mental tests for sleep quality and consciousness monitoring. This will be based on sleep the day before surgery and mini-mental exams before surgery.
  The intraoperative phase Our clinical approach is to admit patients under general anesthesia after regular assessment and monitoring. The following parameters will be recorded intraoperatively.
  After surgery As usual, patients are brought to the PACU after awakening. It will be measured Pittsburghb Sleep Quality Index on 3 days, QoR-15 on the last day, and 3D CAM or ICU-CAM for 3 days postoperatively. Patients will stay in the ward and intensive care unit for 72 hours and be called for 72 hours after release.

SUMMARY:
Background: Delirium is a neurocognitive illness that has lately been connected to sleep difficulties. It is a stressful condition. is still not fully understood. A poor sleep burden and its progress were investigated in this study to determine their correlations with the risk of delirium following surgical procedures.

Methods: Between August 1st and December 5th, 2023, 124 patients undergoing non-cardiac general anesthesia (mean age 63.68 ± 8.81 years [SD]; range 46-82 years) reported on their sleep characteristics. PSQI, 1- sleep duration, 2- sleep disturbance, 3- sleep latency, 4- daytime dysfunction resulting from sleepiness, 5- sleep efficiency, 6- overall sleep quality, and 7- usage of sleep medications were among these sleep characteristics. Seven component scores, ranging from 0 (no difficulty) to 3 (extreme difficulty), are obtained while assessing the PSQI. The global score ranges from 0 to 21 and is calculated by adding the component scores. Higher scores indicate poorer sleep quality. A three-day median follow-up time was used to analyze hospitalization records to gather data on new-onset delirium (n = 26). Approximately 124 people on average, with a mean.

DETAILED DESCRIPTION:
The global old population has grown as life quality has improved. According to WHO and UN publications, people 65 and older are mostly examined, and 60 and older are examined. The Turkish Statistical Institute (TUIK) reports 8 million,245 thousand 124 senior people in Turkey as of December 31, 2022. In December 2021, 9.7% of the population was 65 or older.

In 2021, 9.56% of the global population was 65 or older. Countries' aging processes vary. In 2021, 28.7% of Japan's population was elderly, while the United Arab Emirates had 1.4%. The rate of elderly patients over 65 obtaining general anesthesia for surgery has also grown. Noncardiac surgery often causes delirium in 10-40% of patients. Delirium increases the likelihood of postoperative mortality and poor neurocognitive recovery. The patient, family, and healthcare system are affected by postoperative delirium.

Delirium is difficult to avoid and cure because to its unknown pathophysiology. Evidence suggests that age, frailty, comorbidities, and substance addiction are predisposing and triggering factors. Other risk factors for delirium include perioperative opioid and benzodiazepine usage, operation severity and type, extreme pain, neuroinflammation, and electrolyte problems. Delirium in critically ill individuals is characterized by organ malfunction, acute-onset cognitive impairment, visual hallucinations, delusions, and illusions.

Initial cognitive impairment, acute sickness, dehydration, and aging enhance hospitalized patient delirium. Male gender, alcohol addiction, fractures, depression, visual impairments, and dementia predispose to delirium; restraint, nutritional disorders, multiple medications, urinary catheter, infections, too much or too little sensory stimulation (social isolation), noise, pain, neuroleptics or narcotics, frequent hospital room changes, no clock, no glasses, Surgery, medical procedures, and intensive care can cause delirium (2,16-18).

Critically sick individuals have poor sleep quality and quantity. Sleep disturbances can have a substantial personal and socioeconomic impact on people with respiratory, cardiovascular, metabolic, and mental diseases. In critically ill individuals, severe sleep quality and quantity disruption can cause neurological problems and increased morbidity. After discharge, critically sick individuals may develop acute anxiety and depression due to sleep deprivation.

Melatonin, the pineal gland's major neurohormone, regulates circadian rhythm is anti-inflammatory, antitoxic, hypnotic, anticonvulsive, sedative, and analgesic. Due to noise, 24-hour artificial light, limited natural light, more severe disease severity than general wards, and widespread use of sedative and narcotic drugs, intensive care unit patients' melatonin secretion is severely suppressed. These factors can increase nocturnal wakefulness, shorten sleep, and lower sleep quality. Sleep deprivation alters the sleep-wake cycle, and aberrant melatonin excretion is linked to delirium, a common organ malfunction that affects 45% to 87% of intensive care patients. Delirium is characterized by impaired consciousness with cognitive changes (hyperactive, hypoactive, or mixed) and is associated with longer mechanical ventilation and intensive care time, higher mortality, cognitive sequelae, and higher hospital costs. Sleep deprivation and delirium influence the prefrontal and parietal cortices of the central nervous system, causing neurohormonal alterations such as decreased acetylcholine or increased dopamine. It will be believed sleep can cause delirium.

Because sleep and delirium share processes, this study examines how preoperative sleep quality affects postoperative delirium in over 45 and elderly patients over 65 who receive general anaesthesia. Second, it'll be assessed for postoperative sleep and healing.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if:

  1. Patients receiving general anesthesia
  2. Elective noncardiac surgery lasting more than 2 hours
  3. Patients in the ASA2-3 risk group
  4. Patients aged >45 years

Exclusion Criteria:

* Patients will not be eligible if:

  1. Septic table (clinically diagnosed by the relevant anesthesiologist)
  2. Inadequate recording of delirium assessment;
  3. Previous history of post-surgical delirium
  4. Current or previously diagnosed neurocognitive disease.
  5. Patients who are foreigners or have difficulty communicating due to communication problems.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the sample size analysis, it was determined that there should be 72 patients for each group with an alpha margin of error of 0.05, with a power rate of 80% for comparison of two groups. The effect used for this calculation was calculated as 0.417, and the actual power was calculated as 0.801, based on similar studies. As a result of the analysis, considering the drop out rate, it was planned to include 75 patients for each group.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Sleep quality and delirium index | Preoperative, and post operative period up to 3 days.
  Will be evaluate the relationship between preoperative sleep quality and postoperative delirium.

SECONDARY OUTCOMES:
Preop. and postop. sleep quality index | Preoperative, and post operative period up to 3 days..
  Will be evaluate the effect of preoperative sleep quality on postoperative sleep quality

OTHER OUTCOMES:
Sleep quality and QR 15 score | Preoperative, and post operative period up to 3 days..
  Will be evaluate the effect of preoperative sleep quality on the postoperative recovery process

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Tire, Assoc. Prof., Principal Investigator — Konya City Hospital; Dilek Ateş, MD, Study Director — Konya City Hospital
Locations (1):
- Yasin Tire, Konya, Meram, Turkey (Türkiye)